CLINICAL TRIAL: NCT04563078
Title: Effect of Transcranial Magnetic Stimulation (TMS) on PTSD Neuroimaging and Psychophysiological Biomarkers
Brief Title: Effect of TMS on PTSD Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sanne van Rooij, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000338; K01MH121653 (NIH)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Transcranial Magnetic Stimulation; PTSD; Biomarkers; Neuroimaging; Psychophysiology
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Transcranial Magnetic Stimulation (TMS) (Experimental): TMS is a noninvasive treatment that uses magnetic fields to induce a small electric current in specific brain regions.
  Interventions: Device: Transcranial Magnetic Stimulation (TMS)
- Sham Transcranial Magnetic Stimulation (TMS) (Sham Comparator): Sessions of Sham Transcranial Magnetic Stimulation (TMS) will be conducted.
  Interventions: Procedure: Sham Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS) — 10-day treatment (2 per day with 10 minute break, 20 sessions in total) of active Transcranial Magnetic Stimulation (TMS). TMS is a noninvasive treatment that uses magnetic fields to induce a small electric current in specific brain regions.
  Arms: Transcranial Magnetic Stimulation (TMS)
Procedure: Sham Transcranial Magnetic Stimulation (TMS) — 10-day treatment (2 per day with 10 minute break, 20 sessions in total) of sham control.
  Arms: Sham Transcranial Magnetic Stimulation (TMS)

SUMMARY:
The study will (1) assess feasibility of a TMS treatment in an underserved population; (2) determine if this TMS treatment protocol improves PTSD symptoms and biological markers of PTSD such as brain functioning and startle responses; (3) define new brain targets for future TMS studies; (4) provide the first data for individual differences, which will help personalize treatment for PTSD patients; (5) improve knowledge of the neurobiology of PTSD and treatment response.

DETAILED DESCRIPTION:
Posttraumatic stress disorder is a psychiatric disorder that can develop in response to a traumatic event, and half of civilians living in inner-city areas with high levels of violence suffer from PTSD. The currently recommended treatment for PTSD is focused on discussing the trauma, but a third to half of patients cannot participate or do not benefit from this treatment, especially individuals with low levels of education or literacy. Therefore, new treatments for PTSD are needed.

The study will (1) assess feasibility of a TMS treatment in an underserved population; (2) determine if this TMS treatment protocol improves PTSD symptoms and biological markers of PTSD such as brain functioning and startle responses; (3) define new brain targets for future TMS studies; (4) provide the first data for individual differences, which will help personalize treatment for PTSD patients; (5) improve knowledge of the neurobiology of PTSD and treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age.
* Meet for partial PTSD, defined as 3 out of 4 symptom clusters always including cluster E (alterations in arousal and reactivity) according to the DSM-5 criteria using the Clinician-Administered PTSD Scale (CAPS-5).
* Capable and willing to provide informed consent.
* Able to adhere to the treatment schedule.

Exclusion Criteria:

* Having active suicidal intent or plan as defined by a positive answer to questions 4 and/or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS): Screening version; or in the clinician's opinion, is likely to attempt suicide within the next six months.
* Unstable psychotropic medication status. Participants taking psychotropic medications (i.e.,antidepressants, antipsychotics, benzodiazepines and anticonvulsants, etc.) can be enrolled in the study as long as medication type and dose has been stable for at least 6 weeks, and additionally, medication type or dose does not change during the course of the study.
* Lifetime diagnosis of psychotic disorder or bipolar I disorder per diagnostic interview.
* Diagnosed with the following conditions: a neurological disorder, including a history of seizures, cerebrovascular disease, primary or secondary tumors in CNS, stroke, cerebral aneurysm or movement disorder or any lifetime history of loss of consciousness for more than 5 minutes due to head injury.
* History of cranial surgery, metallic particles in the eye or head (exclusive of mouth), implanted cardiac pacemaker or any intra-cardiac lines, implanted neurostimulators, intra-cranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or implanted medical pumps.
* Current substance abuse or dependence as indicated by a score of 6 or higher on the Drug Abuse Screening Test (DAST).
* Current alcohol abuse or dependence as indicated by a score of 8 or higher on the Alcohol Use Disorder Identification Test (AUDIT).
* Being pregnant or a positive pregnancy test at the beginning of each TMS treatment week for sexually active women of childbearing age who are on reliable birth control.
* Currently participating in another clinical study or enrolled in another clinical study within 30 days prior to this study or started (new) treatment for PTSD within 3 months prior to this study.
* Previously treated with TMS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-09-28 (Actual)

PRIMARY OUTCOMES:
Change in Amygdala Reactivity during fear processing pre- to post-treatment | Baseline, day 10
  Change in Amygdala Reactivity during fear processing pre- to post-treatment will be assessed
Change in skin conductance response to trauma cues pre- to post-treatment | Baseline, day 10
  Change in skin conductance response to trauma cues pre- to post-treatment will be assessed

SECONDARY OUTCOMES:
Change in inhibition-related activation in the ventromedial prefrontal cortex (vmPFC) pre- to post-treatment | Baseline, day 10
  Change in inhibition-related activation in the ventromedial prefrontal cortex (vmPFC) pre- to post-treatment will be assessed
Change in inhibition-related activation in the hippocampus pre- to post-treatment | Baseline, day 10
  Change in inhibition-related activation in the hippocampus pre- to post-treatment will be assessed
Change in ventromedial prefrontal cortex (vmPFC)-amygdala functional connectivity pre- to post-treatment | Baseline, day 10
  Change in vmPFC-amygdala functional connectivity pre- to post-treatment will be assessed
Change in dorsolateral prefrontal cortex (DLPFC)-amygdala functional connectivity pre- to post-treatment | Baseline, day 10
  Change in DLPFC-amygdala functional connectivity pre- to post-treatment will be assessed
Change in Fear-Potentiated Startle Responses to danger and safety cues pre- to post-treatment. | Baseline, day 10
  Change in Fear-Potentiated Startle Responses to danger and safety cues pre- to post-treatment will be assessed
Change in discrimination between danger and safety cues pre- to post-treatment | Baseline, day 10
  Change in discrimination between danger and safety cues pre- to post-treatment will be assessed
Change in Post-traumatic stress disorder (PTSD) hyperarousal symptoms pre- to post-treatment | Baseline, day 10
  Change in PTSD hyperarousal symptoms pre- to post-treatment will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Sanne van Rooij, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT04563078/ICF_001.pdf